CLINICAL TRIAL: NCT02002741
Title: Adding Paracetamol to Ibuprofen for Treatment of Patent Ductus Arteriosus in Preterm Infants: A Pilot, Double Blind, Randomized, Placebo-control Trial
Brief Title: Adding Paracetamol to Ibuprofen for Treatment of Patent Ductus Arteriosus in Preterm Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IBUACA CTIL
Record Dates: First submitted 2013-11-24; First posted 2013-12-06 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Ductus Arteriosus, Patent
Keywords: patent ductus arteriosus; PDA; Preterm; Infant; Electrocardiography; Paracetamol; Acamol; ibuprofen; Placebo
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen + Paracetamol (Active Comparator): Ibuprofen 10mg/kg once --> 5mg/kg twice, q 24h for total of 3 doses
  + Intravenous Paracetamol : Loading dose 20mg/kg --> 10 mg/kg q6h for total of 12 doses
  Interventions: Drug: Paracetamol
- Ibuprofen + Placebo (Placebo Comparator): Ibuprofen 10mg/kg once --> 5mg/kg twice, q 24h for total of 3 doses
  + Placebo (NaCl 0.9%) , Intravenous , at equal volume to the paracetamol in the paracetamol arm, total of 12 doses given q 6h.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — Ibuprofen 3 doses administered q24h + Paracetamol 12 doses administered q 6h
  Other Names: Acetaminophen; Acamol
  Arms: Ibuprofen + Paracetamol
Drug: Placebo — Ibuprofen 3 doses administered q24h + Placebo : 12 doses administered q 6h
  Other Names: NaCl 0.9%
  Arms: Ibuprofen + Placebo

SUMMARY:
The purpose of this study is to determine if adding paracetamol to ibuprofen is superior to ibuprofen only for treatment of patent ductus arteriosus (PDA) in preterm infants.

DETAILED DESCRIPTION:
Randomized control trial to determine if adding paracetamol to ibuprofen is superior to ibuprofen only for treatment of patent ductus arteriosus (PDA) in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at 24-37 gestational age
* diagnosis of Hemodynamically significant patent ductus arteriosus
* Medical staff decided to treat with Ibuprofen
* Parents have signed informed consent

Exclusion Criteria:

* Contraindication for ibuprofen
* Alanine transaminase /Aspartate transaminase≥ 200 U/L
* Significant congenital heart disease

Ages: 2 Days to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of patent ductus arteriosus closure | 3-10 days after first dose of Ibuprofen + study drug
  By echocardiography

SECONDARY OUTCOMES:
Adverse effects | until discharge home (usually within 2-3 months since recruitment)
  Renal and liver function, gastrointestinal complications will be assessed from the patient's medical records
The need for surgical ligation for PDA | 3-21 days after first dose of Ibuprofen + study drug
  need for surgical ligation for PDA

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No